CLINICAL TRIAL: NCT02420925
Title: Effect of Celiac Plexus Block on Gastric Emptying and Symptoms Caused by Gastroparesis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment "0"
Sponsor: Linda Nguyen (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor-Investigator, Linda Nguyen, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: celblockgastro
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Celiac Plexus Block
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Celiac Plexus Block (Experimental): There is one treatment arm who undergoes celiac plexus block.
  Interventions: Procedure: Celiac Plexus Block

INTERVENTIONS:
Procedure: Celiac Plexus Block — Patients will undergo celiac plexus block via upper endoscopy with endoscopic ultrasound guidance. Injections will be performed using 0.75% bupivicaine and 40mg/ml of triamcinolone, ideally 1ml each directly into the celiac ganglia. If no ganglia is identifiable, then the injection will be performed into the celiac space, located at the take off of the celiac artery from the aorta.

SUMMARY:
The investigators hypothesize that in patients with gastroparesis, gastric emptying will improve with celiac plexus block. By improving gastric emptying, symptoms related to gastroparesis including nausea, vomiting, bloating, abdominal pain, and weight loss, will also improve.

In order to study this hypothesis, the investigators will enroll patients with gastroparesis who are non-responsive to the current treatments available. Patients will fill out a questionnaire to assess the severity of their symptoms then undergo Ansar testing (a non-invasive test) to measure their autonomic function respectively. Then, patients will undergo a celiac plexus block which is performed via an upper endoscopy. One week after the procedure, patients will be asked to undergo a gastric emptying study as well as repeat the Ansar testing to evaluate for any improvement in the gastric emptying and autonomic function respectively. Patient will be asked to repeat the questionnaire, one, two, three, and eight weeks after their procedure.

DETAILED DESCRIPTION:
The investigators will identify patients with gastroparesis due to idiopathic causes (including post-viral) and diabetes who have undergone a 4 hour gastric emptying study showing delayed gastric emptying. Patients enrolled must have clinical symptoms due to gastroparesis including nausea, vomiting, abdominal pain, early satiety, bloating, reflux, postprandial fullness or weight loss. Patients included in the study may be refractory to treatment or ineligible for current standard of care with metoclopramide, domperidone, macrolide antibiotics, or pyloric injections with botulinum toxin.

Patients who agree to enroll in the study will sign an informed consent which will explain study purpose along with the risks of the procedures involved in the study. One of the team members will also explain the study to the patient either over the phone or in person and answer any questions they may have in regards to the study.

Patients who are enrolled in the study will fill out a questionnaire comprised of the gastroparesis cardinal symptom index daily diary (GCSI-DD) and visual analog scale (VAS) to assess severity of nausea, vomiting, abdominal pain, and bloating. Then, patients will undergo autonomic function measurements using the Ansar system which is a non-invasive measurement of the autonomic system using blood pressure, heart rate, and respiratory rate monitoring. Ansar testing takes approximately 15 minutes.

Subsequently, patients will undergo a celiac plexus block, performed endoscopically with EUS- guidance by Ann Chen. Injections will be performed using 0.75% bupivicaine and 40mg/ml of triamcinolone, ideally 1ml each directly into the celiac ganglia. If no ganglia is identifiable, then the injection will be performed into the celiac space, located at the take off of the celiac artery from the aorta. One week after their block, a gastric emptying study and Ansar testing will be performed. The GCSI-DD/VAS questionnaire will be repeated 1 week, 2 weeks, 3 weeks, and 2 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have gastroparesis due to idiopathic causes (including post-viral) and diabetes who have undergone a 4 hour gastric emptying study showing delayed gastric emptying
* Patients may have been or currently on therapy for their gastroparesis including metoclopramide, domperidone, macrolide antibiotics, sapropterin dihydrochloride, or pyloric botox injections can be included
* Patients who have undergone placement of electrical gastric stimulator >6 months after enrollment can be included

Exclusion Criteria:

* Patients with suspected mechanical obstruction resulting in delayed gastric emptying, patients chronically using narcotics (>3 times per week)
* Patients who have undergone placement of gastric electrical stimulation device within 6 months of enrollment.
* Patients with any history of small bowel obstruction and major abdominal surgeries (excluding appendectomy, cholecystectomy, Nissen fundoplication, or pelvic surgeries).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Increased gastric emptying | One week after intervention
  We will assess for increased gastric emptying via a SmartPill study, one week after celiac plexus block is performed.
Improvement of gastroparesis based on GCSI-DD score | 2 months
  One, two, three weeks after the procedure as well as 2 months after the celiac plexus block, the patients will fill out a questionnaire questionnaire comprised of the gastroparesis cardinal symptom index daily diary(GCSI-DD).

SECONDARY OUTCOMES:
Improvement of individual symptoms related to gastroparesis based on VAS score | 1week-2 months after procedure
  One, two, and three weeks after the celiac plexus block as well as 2 months after the procedure, the patients will fill out a VAS questionnaire to assess their symptoms related to their gastroparesis.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Nguyen, MD, Principal Investigator — Stanford University; Irene Sonu, MD, Study Director — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

REFERENCES:
- [Background] Memis D, Inal MT, Temizoz O, Genchallac H, Ozdemir H, Sut N. The effect of celiac plexus block in critically ill patients intolerant of enteral nutrition: a randomized, placebo-controlled study. Anesth Analg. 2010 Apr 1;110(4):1071-5. doi: 10.1213/ANE.0b013e3181cde870. Epub 2010 Jan 26. PMID 20103540 (Retraction: PMID 21106975 Shafer SL. Anesth Analg. 2010 Dec;111(6):1561)